CLINICAL TRIAL: NCT02425956
Title: Non-invasive Quantification of Liver Iron With MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 114-2014-GES-0039
Record Dates: First submitted 2015-03-16; First posted 2015-04-24 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Iron Overload
MeSH Terms: conditions — Iron Overload

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI imaging of liver (Experimental): GE Optima/Discovery® MRI imaging data of the liver and surrounding tissues will be acquired using 1.5T and 3.0T GE Healthcare (GEHC) IDEAL IQ scans and commercially available 1.5T MRI scans conducted according to the FerriScan®
  Interventions: Device: GE Optima/Discovery® MRI data of the liver

INTERVENTIONS:
Device: GE Optima/Discovery® MRI data of the liver — GE Optima 1.5T®/Discovery 3.0T® MRI data scanning data of the liver and surrounding tissues will be acquired using both field strengths for GE IDEAL IQ® and single field strength with FerriScan® (Resondence Health) Specialized Reconstruction Service, according instructions provided by manufacturer
  Other Names: GE Optima/Discovery® MRI; FerriScan® (Resondence Health); GE IDEAL IQ®

SUMMARY:
This study is being conducted to build a library of prospectively collected clinical data from subjects with iron overload examined with commercially available MRI devices. This data library is intended for use in future engineering development and other research activities, including future regulatory submissions.

DETAILED DESCRIPTION:
This study is being conducted to build a library of prospectively collected clinical data from subjects with iron overload examined with commercially available MRI devices. This data library is intended for use in future engineering development and other research activities, including future regulatory submissions. Data from human subjects is required to develop and test Magnetic resonance (MR) reconstruction techniques that can provide quantitative information about tissue properties, such as volumetric fat and iron concentrations. Collection of MR data and corresponding quantitative liver iron concentration (LIC) data is necessary for development of MR techniques that can show both overall and regional iron concentrations of in vivo tissues. These techniques may provide viable alternatives to invasive and expensive conventional liver biopsy and to less accurate serum biomarker testing, potentially benefiting future clinical patients with iron overload.

MR image data and corresponding quantitative data about serum and liver iron levels will be collected from each subject in this study. These datasets are considered suitable for future development and testing of MR reconstruction software, including MR reconstruction algorithms developed by General Electric Healthcare (GEHC) to use Longitudinal relaxation rate equal to the reciprocal of T2 relaxation time (1/T2) (R2) techniques to assess LIC. To achieve a sufficiently diverse library for future testing, MRI data of the liver and surrounding tissues will be acquired using 1.5T and 3.0T GEHC IDEAL IQ scans and commercially available 1.5T MRI scans conducted according to the FerriScan® Specialized Reconstruction Service guidelines (Resonance Health, Claremont, AU). Quantitative hematologic (serum ferritin) based on blood testing and FerriScan® Analysis Service LIC reports will be collected for each subject.

ELIGIBILITY:
Inclusion Criteria

1. Be at least ten (10) years of age;
2. Have clinical history of iron overload;
3. If female of childbearing potential (not surgically sterile or post-menopausal), be determined non-pregnant by the medical co-investigator and/or a delegated physician on the study staff or are demonstrated non-pregnant by negative urine pregnancy test administered within the 24 hour period before participating in study procedures;
4. Provide evidence of willingness to participate by providing written informed consent to participate OR, if aged less than 18 years (<18) be willing to provide written assent to participate and have parent(s) or legal guardian(s) willing to provide written informed consent for the subject's participation;
5. Be able to hear and understand instructions without assistive devices;
6. Have necessary mental capacity to understand instructions be able to comply with protocol requirements;
7. Be able to remain relatively motionless for the expected duration of imaging procedures (maximum of approximately 90 minutes).

Exclusion Criteria

1. Have medical history of present or prior focal liver disease, such as neoplasms or vascular abnormalities;
2. Have contraindication(s) to MRI scanning per the routine MR Safety Screening policy of the investigational site;
3. Are scheduled for surgery, changes in dosage or type of chelating medications, or other medical interventions in between blood draw and MRI scanning that could be expected to impact study results or conduct;
4. Have had or plan to have a change in dosage or type of chelating medications (such as Deferoxamine or Deferasirox) within the 3 days prior to the first study procedure (blood draw or MRI, whichever comes first);
5. Are minor subjects with parent(s) or legal guardian(s) that require that they accompany the subject into the MR environment;
6. Have previously participated in this study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Korosec, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRI Imaging of Liver
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MRI Imaging of Liver
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 15
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Per Subject Evaluable DICOM Data Sets From Liver MRI
Description: The primary outcome measure is collection of evaluable (based on physician determination) MR DICOM datasets including valid 1.5 and 3.0T image data, P-file, R2* maps, and raw data for each enrolled subject. The datasets were gathered via three independent MR scans conducted within a three hour time block, with up to ten minutes break in between.
Time Frame: 48 hours pre or 24 hours post blood draw
Population: MR DICOM datasets were gathered for each enrolled subject (total of three scans per subject equals one complete dataset)
Measure: Count of Participants; unit: Participants
Arm/Group | MRI Imaging of Liver
Number analyzed (Participants) | 21
Participants | 21

2. Secondary Outcome: Serum Ferritin Based on Blood Draw
Description: The secondary outcome is collection of serum ferritin from hematologic analysis (blood draw analyzed by site central lab).
Time Frame: 48 hours post MR scan or 24 hours pre MR scan
Population: Every enrolled subject
Measure: Mean (Standard Deviation); unit: mg FE /g dry
Arm/Group | MRI Imaging of Liver
Number analyzed (Participants) | 21
mg FE /g dry | 8.3 (7.71400705)

ADVERSE EVENTS:
Time Frame: Date collected during duration of study enrollment through completion
Arm/Group | MRI Imaging of Liver
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No